CLINICAL TRIAL: NCT03647995
Title: Probiotics in the Prevention of Antibiotic Induced Diarrhea and Clostridium Difficile Associated Diarrhea; A Randomized Double Blind Placebo Controlled Trial.
Brief Title: Probiotics in the Prevention of Antibiotic Induced Diarrhea and Clostridium Difficile Associated Diarrhea.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Were not able to enroll enough participants due to shortage of study staff
Sponsor: Yara El Helou (Other)
Collaborators: Pharma M (Unknown)
Responsible Party: Sponsor-Investigator, Yara El Helou, Medical Student, Saint-Joseph University
Organization: Saint-Joseph University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ProbioSJU
Record Dates: First submitted 2018-08-23; First posted 2018-08-27 (Actual); Last update posted 2020-10-26 (Actual); Status verified 2020-10

CONDITIONS: Diarrhea, Clostridium Difficile
Keywords: Probiotics; Diarrhea; Clostridium difficile; Antibiotics; Antibiotic-associated diarrhea; Clostridium difficile-associated diarrhea; Microbial flora
MeSH Terms: conditions — Diarrhea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The randomization will be taken care of by the hospital pharmacy which will not be in contact with the patient.
  The intern/resident who will recruit a patient in the study will not be in direct contact with the pharmacy.
  The order will be sent to the pharmacy which, following a randomization sheet, will then send a neutral box containing a probiotic or a placebo product.
  Only once the trial comes to an end, the investigator will receive from the pharmacy the randomization sheet and will then know which patient was given a probiotic and which was given a placebo regimen.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic-receiving group (Active Comparator): The probiotic-receiving group will receive once daily probiotics containing 25Bn CFU of which: 5Bn CFU Lactobacillus rhamnosus GG, 5Bn CFU Sacchromyces boulardii, 5Bn CFU Bifidobacterium breve, 4.5Bn CFU Bifidobacterium lactis, 2.5 Bn CFU Lactobacillus acidophilus, 2.5Bn CFU Lactobacillus plantarum and 500Mn CFU Lactobacillus reuteri.
  Interventions: Dietary Supplement: Probiolife by Green Made (Pharma M)
- Placebo (Placebo Comparator): The placebo group will receive once daily, identical capsules containing 0 Bn CFU.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Probiolife by Green Made (Pharma M) — A box containing 30 capsules of a dietary supplement containing 25 Bn CFU (detailed in previous sections)
  Arms: Probiotic-receiving group
Other: Placebo — A box containing 30 capsules containing an inactive substance with 0 Bn CFU.
  Arms: Placebo

SUMMARY:
The objective of this study is to determine the efficacy of probiotics containing 25Bn (billion) CFU (colony-forming unit) of Lactobacillus rhamnosus, Sacchromyces boulardii and Bifidobacterium breve in the prevention of antibiotic induced diarrhea and Clostridium difficile diarrhea.

The chosen population consists of 190 hospitalized patients taking antibiotics. Preselected and randomized patients will take probiotics once daily until 1 week after the course of antibiotic is over or a placebo with 0 CFU.

The primary outcome is to detect the occurrence of an antibiotic-associated diarrhea. The secondary outcome is to assess the presence of Clostridium difficile toxins in stool culture.

DETAILED DESCRIPTION:
Antibiotic-associated diarrhea (AAD) and Clostridium difficile associated diarrhea (CDAD) are a common nosocomial complication following antibiotic use. AAD and CDAD are most importantly associated with an increase in morbidity and mortality -especially in the elderly population- thus also contributing to a significant financial burden.

It was reported that 5-25% of patients on antibiotics will develop an AAD of which 10-20% are caused by Clostridium difficile. Furthermore, the widespread use of broad spectrum antibiotics is contributing to the increased incidence of CDAD.

The adult human intestinal tract contains up to 100 trillion micro-organisms. This microbiota is essential and injury to this barrier can result in multiple GI diseases such as infection by pathogens.

Probiotics are defined as "live micro-organisms which when administered in adequate amounts confer a health benefit on the host" [WHO 2007]. Many studies suggest that the use of probiotics and probiotic containing milks will significantly decrease the risk of AAD and maybe even CDAD.

This study is a randomized double-blind, placebo controlled trial using probiotics containing 25 Bn (billion) CFU of which: 5Bn CFU Lactobacillus rhamnosus, 5Bn CFU Sacchromyces boulardii, 5Bn CFU Bifidobacterium breve, 4.5Bn CFU Bifidobacterium lactis, 2.5 Bn CFU Lactobacillus acidophilus, 2.5Bn CFU Lactobacillus plantarum and 500Mn (million) CFU Lactobacillus reuters or a placebo containing 0 CFU in order to assess the role of probiotics in the prevention of AAD and CDAD.

Diarrhea is defined as more than two liquid stools for a period greater than 3 days and which is considered by the patient as an increase in stool quantity compared to regular basis. This issue will be recorded by the intern/resident. However; if the patient starts his antibiotic regimen in the hospital and is later discharged at home; the patient will be kept in direct contact with a specific intern/resident and will inform him of the presence of diarrhea.

The presence of Clostridium Difficile Toxins A and/or B while on antibiotics and for a month after that will be assessed in the context of diarrhea in hospitalized patients only.

Our patients will be recruited from Hotel-Dieu de France hospital. This includes patients of all ages who are prescribed antibiotics (single or multiple; oral or IV) assuming that they are able to eat/drink so that they can take the probiotic pills.

Patients also need to be able to sign a consent form by themselves.

Both groups (probiotic and placebo) will begin treatment within a maximum of 48 hours after the start of the antibiotic regimen and for the entire duration of antibiotic therapy. This regimen will be continued a week after the antibiotic therapy is stopped. Researchers will verify patients' compliance on a daily basis in the hospital and on a weekly basis once the patient is discharged.

The exclusion criteria are the following: diarrhea on admission; bowel pathology that could result in diarrhea (eg. IBD), bowel surgeries and pouches; immunocompromised state (including febrile aplasia, immunosuppressive therapy, ICU patients, HIV-positive patients and renal transplant patients); prosthetic heart valves or history of endocarditis and rheumatic heart disease; use of metronidazole, vancomycin or fidaxomycin prior to stool culture for Clostridium difficile toxins.

Via our computerized medical system, investigators will be able to identify patients who start an antibiotic regimen. Those who match the trial's inclusion and exclusion criteria will be included in the trial after a written consent form is obtained.

The hospital pharmacy will provide them with probiotic or placebo boxes each containing 30 capsules that look similar.

Once the antibiotic regimen is finished, the probiotic/placebo course is continued for another week with a final follow up 4 weeks after the last course of antibiotics. If the patient is discharged before the end of his antibiotic course, he will be given enough probiotics/placebo until the end of his antibiotic course and for a week after that. Those patients will be followed with a weekly phone call and a final follow up 4 weeks after the last course of antibiotics.

If the patient presents with diarrhea in the hospital, a stool sample will be collected to check for Clostridium Difficile Toxins A and B.

If these cultures come back positive, the probiotic/placebo regimen is then stopped.

In order to detect an absolute difference of 20% between the proportion of patients in the placebo group with AAD (considered 30%) and the probiotic group (considered 10%) with α=0.05 and a power of 90% we estimated that we needed a sample size of 164 (82 in each group). Researchers furthermore considered a 10% risk of loss of contact with the patient and therefore estimated a sample size of 180 (90 in each group).

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized on antibiotics (single or multiple; oral or IV) assuming that they are able to eat/drink so that they can take the pills.
* Regimen started within 48 hours of first course of antibiotics.
* Able to sign a consent form.

Exclusion Criteria:

diarrhea on admission; bowel pathology that could result in diarrhea (eg. IBD), bowel surgeries and pouches; immunocompromised state (including febrile aplasia, immunosuppressive therapy, ICU patients, HIV-positive patients and renal transplant patients); prosthetic heart valves or history of endocarditis and rheumatic heart disease; use of metronidazole, vancomycin or fidaxomycin prior to stool culture for Clostridium difficile toxins.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-02-02 (Actual); Study Completion 2019-02-02 (Actual)

PRIMARY OUTCOMES:
Occurrence of an antibiotic-associated diarrhea. | From the first day of inclusion in the trial up to a month after the antibiotic regimen is stopped.
  Diarrhea is defined as more than two liquid stools for a period greater than 3 days and which is considered by the patient as an increase in stool quantity compared to regular basis, evaluated in a patient on antibiotics.

SECONDARY OUTCOMES:
Presence of Clostridium difficile toxins in stool culture. | Upon eventual onset of diarrhea, from the first day of inclusion in the trial and up to a month after the antibiotic regimen is stopped; in hospitalized patients only.
  Presence of Clostridium difficile toxins A and/or toxins B in the stool culture, evaluated in a patient on antibiotics presenting with diarrhea.

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Joseph University of Beirut, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No